CLINICAL TRIAL: NCT06182553
Title: Effect of Expiratory Rib Cage Compression and/or PEEP-ZEEP Maneuver on Oxygenation, Ventilation, and Airway Secretions Removal in Mechanically Ventilated Patients
Brief Title: Effect of ERCC and/or PEEP-ZEEP Maneuver on Oxygenation, Ventilation, and Airway Secretions Removal in MV Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Damanhour University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MV Patients
Record Dates: First submitted 2023-11-26; First posted 2023-12-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Mechanically Ventilated Patients

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial with four parallel groups will be used in the current study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group (1) : ERCC Group (Experimental): - The researcher will implement the ERCC technique for 10 minutes as follows: the researcher will use both hands bilaterally to gradually squeeze the rib cage (on the anterolateral region of the chest at the level of the last six ribs) in conjunction with chest-wall vibration during the expiratory phase of the ventilatory cycle. From the end of inspiration to the end of expiration, an attempt will be made to compress the rib cage over the region of the lungs that is most affected and the force will be applied every 2 breaths only during the expiration, synchronizing the maneuver rate with the breathing frequency of the subject. At the end of each expiratory phase, rib-cage compression is interrupted to permit free manual hyperinflation-induced inspiration. The ERCC technique will be implemented twice per day.
  Interventions: Other: Expiratory Rib Cage Compression
- Group (2) : PEEP-ZEEP Group (Experimental): * The researcher in the presence of the attending physician will apply the PEEP-ZEEP maneuver in the following manner: During the inspiration phase of the ventilatory cycle, it is proposed to increase PEEP to 15 cmH2O, while maintaining a PIP of 40 cmH2O. Following the completion of five ventilatory cycles, PEEP will be abruptly decreased to 0 cmH2O during the expiration phase, referred to as ZEEP. Subsequently, during the subsequent inspiration phase, PEEP will be restored to the previously established levels. The maneuver will be repeated for a duration of 10 minutes, with a gap of two ventilatory cycles between every repetition.The PEEP-ZEEP maneuver will be implemented twice per day. At the end of the PEEP-ZEEP maneuver, the patient will receive tracheal suction as mentioned before.
  * The patients will be monitored continuously, and the maneuver will be interrupted if the patients become hemodynamically unstable or develop psychomotor agitation.
  Interventions: Other: PEEP-ZEEP Maneuver
- Group (3) : ERCC + PEEP-ZEEP Group (Experimental): The ERCC technique will be applied as mentioned above, followed by PEEP-ZEEP maneuvers according to the standard steps mentioned before. Also, the patients will be monitored continuously, and the maneuver will be interrupted if the patients become hemodynamically unstable or develop psychomotor agitation.
  Interventions: Other: ERCC + PEEP-ZEEP maneuver
- Group (4) : control Group (No Intervention): * The researcher will observe the conventional nursing care provided by CCNs in the study settings which may affect oxygenation, ventilation, and airway clearance for 30 minutes twice daily for five consecutive days. These conventional nursing practices may include enteral feeding, changing patients' positions, routine suctioning, and other traditional physiotherapies such as chest percussion and vibration.
  * Part II of tool one will be used to assess physiological parameters, and tool two will be used to assess oxygenation, ventilation parameters, and airway clearance indicators for patients in the control group twice per day from the 1st day to the 5th day of the study pre and post-conventional nursing care.

INTERVENTIONS:
Other: Expiratory Rib Cage Compression — Expiratory rib cage compression (ERCC) In this study, ERCC is a technique consisting of bilateral manual compression of the lower rib cage (anterolateral region of the chest at the level of the six last ribs) gradually during the expiratory phase of the ventilatory cycle and release from the compression at the end of the expiration.
  Arms: Group (1) : ERCC Group
Other: PEEP-ZEEP Maneuver — PEEP-ZEEP maneuver In this study, PEEP-ZEEP maneuver refers to PEEP which stands for positive end-expiratory pressure, and ZEEP which stands for zero end-expiratory pressure. In this maneuver PEEP will be incremented to 15 cmH2O throughout five consecutive respiratory cycles, then immediately after the inspiratory phase of the fifth cycle has been ended ZEEP should be done by abruptly reducing PEEP value to 0 cmH2O. The PEEP-ZEEP maneuver should be performed in two sets, consisting of a total of 10 consecutive breathing cycles. Subsequently, the patient is ventilated according to his/her baseline ventilator parameters.
  Arms: Group (2) : PEEP-ZEEP Group
Other: ERCC + PEEP-ZEEP maneuver — - The ERCC technique will be applied as mentioned above, then followed by PEEP-ZEEP maneuvers according to the standard steps mentioned before.
  Arms: Group (3) : ERCC + PEEP-ZEEP Group

SUMMARY:
Mechanical ventilation (MV) is crucial in managing respiratory insufficiency. However, prolonged use can cause complications. Various strategies have been explored to optimize patient outcomes.

Patients receiving IMV face multiple challenges in clearing lung secretions, such as inadequate humidification, high oxygen fractions, use of sedatives/analgesics, basal lung disease, and mechanical interference with secretion elimination near the trachea. Airway suctioning may not be sufficient in clearing the airway of mechanically ventilated patients, especially if they are paralyzed or lack a preserved cough reflex. This can lead to secretion retention, which may cause hypoxemia, atelectasis, ventilator-associated pneumonia, and delay weaning from MV. Bronchial hygiene is believed to improve respiratory system compliance by increasing Cdyn and Cst.

Airway clearance techniques are commonly used in the treatment of patients with IMV to improve their pulmonary function through bronchial clearance, expansion of collapsed lung areas, and balancing of the ventilation/perfusion ratio. Physiotherapy methods including postural drainage, manual rib-cage compression (MRC), manual hyperinflation, positive end-expiratory pressure-zero end-expiratory pressure (PEEP-ZEEP) maneuver, and tracheal suctioning can alleviate atelectasis and improve bronchial hygiene.

Two effective techniques for improving lung function and gas exchange are Expiratory Rib Cage Compression (ERCC) and the PEEP-ZEEP maneuver. ERCC applies external pressure during expiration, and PEEP-ZEEP temporarily reduces Positive End-Expiratory Pressure (PEEP) to 0 cmH2O, followed by a rapid return to the original PEEP level during expiration. Both techniques help to mobilize and remove airway secretions, ultimately improving lung function and gas exchange.

DETAILED DESCRIPTION:
Expiratory rib cage compression is a form of chest physiotherapy that involves squeezing the chest with the hands during expiration and releasing it at the end of expiration to aid in the mobilization of lung secretions, facilitate comfortable inspiration, and promote alveolar ventilation. The concept of manual chest compression was first explored in the 1950s, when Opie et al. proposed that local chest compression produces a "toothpaste" effect, which helps to expel the retained material through the bronchus. This phenomenon piqued the interest of other researchers, leading to a better understanding of the functioning of the mucous layer and the development of therapeutic strategies to improve it.

This technique increases forced expiratory volume by 30% and leads to the resting of the expiratory muscles. Most of all, the technique is quite safe, as it has been employed in some patients for more than 3 years with no complications. Therefore, this technique can be used before the patients' endotracheal suctioning interventions, and it is widely used with mechanically ventilated patients to prevent and/or to treat atelectasis. In addition, removing secretion is essential because accumulated secretions intervene in gas exchange and may delay recovery; coughing can be initiated voluntarily or by reflex.

The positive end-expiratory pressure-zero end-expiratory pressure maneuver considers that by raising PEEP to 15 cmH2O during five cycles, followed by an abrupt reduction of PEEP to 0 cmH2O, gas redistribution occurs through collateral ventilation. Subsequently, small airways are opened, and the adhered mucus is displaced. With the reduction of PEEP, the expiratory flow pattern is modified, causing the secretions located in smaller airways to be transported to the central airways.

While many studies have looked at the effects of rib cage compression (RCC) or the PEEP-ZEEP maneuver individually, there is a need for comparative studies that directly compare these two techniques. Understanding the different effects of these interventions on oxygenation, ventilation, and airway-secretion removal can help critical care nurses (CCNs) choose the most effective strategy for mechanically ventilated patients. Therefore, the purpose of this study is to compare the effects of RCC and the PEEP-ZEEP maneuver on oxygenation, ventilation, and airway-secretion removal in mechanically ventilated patients. By evaluating these outcomes, we can gain insights into the potential benefits and limitations of each technique, ultimately contributing to the optimization of respiratory support strategies in critically ill patients.

The findings of this study can have important implications for CCN clinical practice as they can inform CCNs about the efficacy and safety of RCC and the PEEP-ZEEP maneuver. Improving oxygenation, ventilation, and airway-secretion removal in mechanically ventilated patients can lead to enhanced patient outcomes, reduced complications, and potentially shorter durations of mechanical ventilation and intensive care unit stays.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are aged ≥18 years.
* Patients who have tracheal intubation and are likely to require MV for ≥72 hours.
* Patients who are hemodynamically stable: Heart rate (HR): ≥ 60 b or ≤100 b/min, mean arterial pressure (MAP) ≥ 90 mmHg, central venous pressure ≥ 3 or ≤ 8 cmH2O.

Exclusion Criteria:

* Patients with pneumothorax, rib fracture, and subcutaneous emphysema.
* Patients with traumatic brain injuries and spinal cord injuries.
* Patients with ARDS who require high PEEP levels (>10 cmH2O).
* Patients admitted with pneumonia.
* Pregnant patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
oxygenation | (T0) pre-intervention, (T1) immediately after the intervention, and (T3) up to 30 minutes
  partial pressure of oxygen tension (PaO2). (mmHg) Arterial oxygen saturation (SaO2). (100%) PaO2/FiO2 ratio, and oxygenation index (OI). (mmHg)
ventilation | (T0) pre-intervention, (T1) immediately after the intervention, and (T3) up to 30 minutes
  The partial pressure of carbon dioxide (PaCO2). (mmHg) Tidal volume (Vt). (ml) Positive end-expiratory pressure (PEEP). (CmH2O) Peak inspiratory pressure (PIP). (CmH2O) Minute ventilation (Mv). (L/m) Inspiratory: Expiratory Ratio (I: E ratio). Friction of inspired Oxygen (FIO2). (100%) Pressure Support (PS). (CmH2O) Plateau Pressure (Ppt). (CmH2O) Oxygen flow rate. (L/m) Static compliance (Cst) and dynamic compliance (Cdyn). (L/CmH2O) Respiratory system resistance (Rsr). (CmH2O/L /Sec) Rapid shallow breathing index (RSBI). (Breath /m/L)
airway-secretion removal | (T0) pre-intervention, (T1) immediately after the intervention, and (T3) up to 30 minutes
  1. Oxygenic parameters for airway clearance, such as SpO2 (100%) and end tidal carbon dioxide (ETCO2) (mmHg).
  2. Sputum parameters that include volume (ml), colour, consistency of respiratory secretions cleared from the airways, and frequency of sputum suctioning.
  3. Lung function parameters such as peak inspiratory flow (PIF) (L/m), peak expiratory flow (PEF) (L/m): PIF ratio, peak airway pressure-plateau pressure gradient during constant flow ventilation (CmH2O), respiratory rate (RR) (b/m), maximum airway pressure (CmH2O), and vital capacity (L).
  4. Ventilator graphs, especially flow-volume loops.
  5. Lung sound auscultation (presence or absence of chest crepitations).

SECONDARY OUTCOMES:
duration of mechanical ventilation (days) | 5 days
  effect of ERCC and/or PEEP-ZEEP maneuvers on duration of mechanical ventilation (days)
length of ICU stay (days) | from day 1 till discharge
  effect of ERCC and/or PEEP-ZEEP maneuvers on length of ICU stay (days).

CONTACTS AND LOCATIONS:
Overall Officials: Sahar Younes Othman, ASS-PROF, Study Director — Damanhour University

REFERENCES:
- [Result] Unoki T, Kawasaki Y, Mizutani T, Fujino Y, Yanagisawa Y, Ishimatsu S, Tamura F, Toyooka H. Effects of expiratory rib-cage compression on oxygenation, ventilation, and airway-secretion removal in patients receiving mechanical ventilation. Respir Care. 2005 Nov;50(11):1430-7. PMID 16253149
- [Result] Borges LF, Saraiva MS, Saraiva MAS, Macagnan FE, Kessler A. Expiratory rib cage compression in mechanically ventilated adults: systematic review with meta-analysis. Rev Bras Ter Intensiva. 2017 Jan-Mar;29(1):96-104. doi: 10.5935/0103-507X.20170014. PMID 28444078
- [Result] Zhang J, Wang X, Xie J, Shen L, Mo G, Xie L. Effects of THE PEEP-ZEEP Maneuver in Adults Receiving Mechanical Ventilation: A Systematic Review with Meta-Analysis. Heart Lung. 2024 Jan-Feb;63:159-166. doi: 10.1016/j.hrtlng.2023.10.010. Epub 2023 Nov 2. PMID 37922664
- [Result] Amaral BLR, de Figueiredo AB, Lorena DM, Oliveira ACO, Carvalho NC, Volpe MS. Effects of ventilation mode and manual chest compression on flow bias during the positive end- and zero end-expiratory pressure manoeuvre in mechanically ventilated patients: a randomised crossover trial. Physiotherapy. 2020 Mar;106:145-153. doi: 10.1016/j.physio.2018.12.007. Epub 2019 Feb 3. PMID 30979507
- [Result] de Oliveira TF, Peringer VS, Forgiarini Junior LA, Eibel B. PEEP-ZEEP Compared with Bag Squeezing and Chest Compression in Mechanically Ventilated Cardiac Patients: Randomized Crossover Clinical Trial. Int J Environ Res Public Health. 2023 Feb 5;20(4):2824. doi: 10.3390/ijerph20042824. PMID 36833521
- [Result] Herbst-Rodrigues MV, Carvalho VO, Auler JO Jr, Feltrim MI. PEEP-ZEEP technique: cardiorespiratory repercussions in mechanically ventilated patients submitted to a coronary artery bypass graft surgery. J Cardiothorac Surg. 2011 Sep 13;6:108. doi: 10.1186/1749-8090-6-108. PMID 21914178
- [Result] Santos FR, Schneider Junior LC, Forgiarini Junior LA, Veronezi J. Effects of manual rib-cage compression versus PEEP-ZEEP maneuver on respiratory system compliance and oxygenation in patients receiving mechanical ventilation. Rev Bras Ter Intensiva. 2009 Jun;21(2):155-61. English, Portuguese. PMID 25303345
- [Result] Volpe MS, Guimaraes FS, Morais CC. Airway Clearance Techniques for Mechanically Ventilated Patients: Insights for Optimization. Respir Care. 2020 Aug;65(8):1174-1188. doi: 10.4187/respcare.07904. PMID 32712584
- [Result] Oliveira ACO, Lorena DM, Gomes LC, Amaral BLR, Volpe MS. Effects of manual chest compression on expiratory flow bias during the positive end-expiratory pressure-zero end-expiratory pressure maneuver in patients on mechanical ventilation. J Bras Pneumol. 2019 Mar 11;45(3):e20180058. doi: 10.1590/1806-3713/e20180058. PMID 30864618
- [Result] Dyhr T, Laursen N, Larsson A. Effects of lung recruitment maneuver and positive end-expiratory pressure on lung volume, respiratory mechanics and alveolar gas mixing in patients ventilated after cardiac surgery. Acta Anaesthesiol Scand. 2002 Jul;46(6):717-25. doi: 10.1034/j.1399-6576.2002.460615.x. PMID 12059898
- [Result] Guimaraes FS, Lopes AJ, Constantino SS, Lima JC, Canuto P, de Menezes SL. Expiratory rib cage Compression in mechanically ventilated subjects: a randomized crossover trial [corrected]. Respir Care. 2014 May;59(5):678-85. doi: 10.4187/respcare.02587. Epub 2013 Oct 8. PMID 24106324
- [Result] Unoki T, Mizutani T, Toyooka H. Effects of expiratory rib cage compression and/or prone position on oxygenation and ventilation in mechanically ventilated rabbits with induced atelectasis. Respir Care. 2003 Aug;48(8):754-62. PMID 12890295
- [Result] Bousarri MP, Shirvani Y, Agha-Hassan-Kashani S, Nasab NM. The effect of expiratory rib cage compression before endotracheal suctioning on the vital signs in patients under mechanical ventilation. Iran J Nurs Midwifery Res. 2014 May;19(3):285-9. PMID 24949068
- [Result] Jalil Y, Damiani LF, Basoalto R, Bachmman MC, Bruhn A. A deep look into the rib cage compression technique in mechanically ventilated patients: a narrative review. Rev Bras Ter Intensiva. 2022 Jan-Mar;34(1):176-184. doi: 10.5935/0103-507X.20220012-pt. PMID 35766667
- [Result] Van der Touw T, Mudaliar Y, Nayyar V. Cardiorespiratory effects of manually compressing the rib cage during tidal expiration in mechanically ventilated patients recovering from acute severe asthma. Crit Care Med. 1998 Aug;26(8):1361-7. doi: 10.1097/00003246-199808000-00021. PMID 9710095
- [Result] Hosoe T, Tanaka T, Hamasaki H, Nonoyama K. Effect of positioning and expiratory rib-cage compression on atelectasis in a patient who required prolonged mechanical ventilation: a case report. J Med Case Rep. 2022 Jun 23;16(1):265. doi: 10.1186/s13256-022-03389-5. PMID 35739590
- [Result] Kohan M, Mohammad-Taheri N. Expiratory rib cage compression, endotracheal suctioning, and vital signs. Iran J Nurs Midwifery Res. 2016 May-Jun;21(3):343. doi: 10.4103/1735-9066.180383. No abstract available. PMID 27186215
- [Result] Berti JS, Tonon E, Ronchi CF, Berti HW, Stefano LM, Gut AL, Padovani CR, Ferreira AL. Manual hyperinflation combined with expiratory rib cage compression for reduction of length of ICU stay in critically ill patients on mechanical ventilation. J Bras Pneumol. 2012 Jul-Aug;38(4):477-86. doi: 10.1590/s1806-37132012000400010. English, Portuguese. PMID 22964932
- [Result] Mase K, Yamamoto K, Murakami S, Kihara K, Matsushita K, Nozoe M, Takashima S. Changes in ventilation mechanics during expiratory rib cage compression in healthy males. J Phys Ther Sci. 2018 Jun;30(6):820-824. doi: 10.1589/jpts.30.820. Epub 2018 Jun 12. PMID 29950772
- [Result] Ntoumenopoulos G. Expiratory rib-cage compression, airway suctioning, and atelectasis. Respir Care. 2005 Mar;50(3):387; author reply 387-8. No abstract available. PMID 15779155
- [Result] Ouchi A, Sakuramoto H, Unoki T, Yoshino Y, Hosino H, Koyama Y, Enomoto Y, Shimojo N, Mizutani T, Inoue Y. Effects of Manual Rib Cage Compressions on Mucus Clearance in Mechanically Ventilated Pigs. Respir Care. 2020 Aug;65(8):1135-1140. doi: 10.4187/respcare.07249. Epub 2020 Feb 11. PMID 32047123
- [Result] Morino A, Shida M, Tanaka M, Sato K, Seko T, Ito S, Ogawa S, Takahashi N. Comparison of changes in tidal volume associated with expiratory rib cage compression and expiratory abdominal compression in patients on prolonged mechanical ventilation. J Phys Ther Sci. 2015 Jul;27(7):2253-6. doi: 10.1589/jpts.27.2253. Epub 2015 Jul 22. PMID 26311963
- [Result] D'Angelo E, Miserocchi G, Agostoni E. Effect of rib cage or abdomen compression at iso-lung volume on breathing pattern. Respir Physiol. 1976 Nov;28(2):161-77. doi: 10.1016/0034-5687(76)90036-0. PMID 1070768